CLINICAL TRIAL: NCT02629055
Title: EMG Measurements of Respiratory Muscles for the Titration of Nocturnal Non-invasive Ventilation in Stable Chronic Obstructive Pulmonary Disease Patients: A Randomized Controlled Trial
Brief Title: Respiratory EMG for NIV Titration in Stable COPD Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment during the predefined time frame for the study
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marieke Duiverman, Dr., University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015/383
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Non-invasive ventilation; Respiratory electromyography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Respiratory EMG (Experimental): Additional EMG measurements whilst on NIV will be used to guide the titration of NIV.
  Interventions: Other: Respiratory EMG
- Care as usual (No Intervention): NIV will be initiated according to standard care protocol.

INTERVENTIONS:
Other: Respiratory EMG — Titration of non-invasive ventilation on surface respiratory muscle activity
  Arms: Respiratory EMG

SUMMARY:
The aim of the present study is to investigate whether additional titration on surface electromyography (EMG) of the diaphragm and intercostal muscles improves the outcome of chronic non-invasive ventilation in patients with COPD and stable chronic hypercapnic respiratory failure in terms of better gas exchange after six weeks, lung function, patient comfort and compliance, and less patient ventilator asynchrony. Therefore, the investigators set up a randomized, two-armed crossover trial comparing regular titration with additional respiratory EMG titration of NIV.

DETAILED DESCRIPTION:
Rationale:

Long-term application of nocturnal non-invasive ventilation (NIV) in stable hypercapnic chronic obstructive pulmonary disease (COPD) patients has long been controversial as study results were not unequivocal. However, in the past 7 years, with a change in ventilatory strategy, clear benefits of chronic NIV have been shown in COPD patients with chronic hypercapnic respiratory failure (CHRF), though only in stable disease. As a consequence, this so called high-intensity NIV, which is the concept of using higher positive inspiratory airway pressures (IPAP) levels than used in most of the older trials in addition to controlled ventilation with higher backup breathing frequencies aiming for maximal arterial carbon dioxide (PaCO2) reduction, has gained increasing attention.

However, it is unknown how high-intensity NIV works, and how to titrate the optimal IPAP and optimal backup breathing frequency. Measuring respiratory muscle activity might be a way to titrate NIV in COPD.

Objective:

The aim of the present study is to investigate whether additional titration on surface electromyography (EMG) of the diaphragm and intercostal muscles improves outcomes of chronic NIV in patients with COPD and stable CHRF in terms of better gas exchange after six weeks, lung function, patient comfort and compliance and less patient-ventilator asynchrony (PVA).

Study design:

A randomized, two-armed, crossover trial comparing regular titration with additional respiratory EMG titration of NIV in stable hypercapnic COPD.

One group will be initiated on NIV according to standard care protocol. For the other group, additional EMG measures whilst on NIV will be made to titrate NIV.

Protocol Regular NIV-set up (both groups) Subjects are initiated on NIV according to our own local treatment protocol. NIV is initiated by a registered nurse of our home mechanical ventilation (HMV) centre. Effectiveness is measured with transcutaneous measurements of carbon dioxide (PtCO2).

NIV is supplied through a pressure cycled ventilator, applying both inspiratory airway pressure and expiratory airway pressure to the patient (BiPAP; Synchrony, Respironics, incorporated., Murrysville, USA). A nasal or full face mask (Mirage mask, ResMed Ltd, UK) of proper size is used. The ventilator is set in a spontaneous/ time mode (S/T), with a backup frequency. If needed O2 was added to obtain a saturation of ≥ 90%. A humidifier (HC 150 Fisher & Paykel Healthcare, Australia) is used if needed. In general, the nurse aims to reach a setting with high inspiratory pressures and a moderate breathing backup frequency, with good patient comfort.

Start of the study Patients will be included in the study once they is used to the mask, can sleep at least 6 hours with the ventilator and settings are set as is usual in daily clinical practice. This means that the initial NIV settings are optimized according to the results of an overnight PtCO2 and patient comfort. In daily practice, the specialized nurses of the HMV centre already aim to increase the inspiratory pressure to the highest pressure that is still comfortable for the patient, so that all patients will already be at their highest tolerable pressure.

Once patients agree to participate, a 15-minute EMG measurement is done in all patients while they are ventilated with the settings at that particular moment. Furthermore, patients are asked to complete the severe respiratory insufficiency (SRI) questionnaire.

In the "nurse titrated NIV" group, no additional changes are made to the ventilatory settings. In the "EMG titrated NIV" group, after a 15-minute EMG with the ventilatory settings set by the nurse, the nurse will decrease the backup breathing frequency set by the ventilator by steps of 2 breaths/min to 8 breaths/min (to achieve a pressure support mode of ventilation (completely triggered by the patient)) and then again up to a frequency 2 breaths/min above their spontaneous breathing frequency while on the ventilator (to achieve a controlled mode of ventilation). Each frequency will be measured for 10 minutes, so that the total titration will take about 60-80 minutes. EMG measurements will be done throughout the whole session and will be analyzed the same day. Then, the setting is chosen with the lowest EMG activity and least PVA. The next night an EMG measurement is performed at the chosen setting.

6 weeks After 6 weeks, the overnight EMG measurement is repeated in all patients. Furthermore, a nocturnal PtCO2 measurement is performed, patients are asked to rate how comfortable the patient is with the settings and are asked to fill in the SRI, lung function is assessed and the number of hours use per night is read from the ventilator counting reading. After these measurements are performed, patients are directed to the other titration arm. In patients initially titrated by the nurse, an EMG frequency titration is performed as described above. In the patients initially titrated additionally on the EMG, the investigators will reset the ventilator to the settings applied by the nurse initially.

12 weeks After 12 weeks, the nocturnal EMG measurement, the nocturnal transcutaneous CO2 measurement, the comfort score, the SRI, lung function assessment and compliance rating are repeated in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD) Global initiative of chronic Obstructive Lung Diseases (GOLD) stage III or IV (FEV1 <50 % predicted, FEV1/forced expiratory volume (FVC) < 70% predicted)
* Indication for the initiation of chronic NIV: PaCO2 >6.0 kilopascal (kPa) at rest during daytime.
* Stable COPD (pH >7.35, no exacerbation in the past two weeks)
* Age >18 years

Exclusion Criteria:

* Respiratory insufficiency of any other cause.
* Already initiated on chronic NIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Nocturnal gas exchange (PCO2 (kPa)) | 6 weeks
  PCO2 will be assessed with transcutaneous measurements (TOSCA, Linde Medical Sensors AG, Basel)

SECONDARY OUTCOMES:
Patient comfort measured with a Visual Analogue Scale | 6 weeks
  comfort with NIV setting, measured with a Visual Analogue Scale
Health related quality of life measured with the Severe Respiratory Insufficiency (SRI) questionaire | 6 weeks
  Measured with the Severe Respiratory Insufficiency (SRI) questionaire
Lung volumes | 6 weeks
  Total Lung Capacity (liters) and Residual Volume (liters))
Respiratory muscle strength | 6 weeks
  Maximal inspiratory pressure (kPa)).
Patient-Ventilator Asynchrony (PVA) | 6 weeks
  The investigators will assess PVA's by simultaneously comparing EMG recordings with pressure waves delivered by the ventilator. PVA's are measured as a percentage of the total number of delivered breaths

CONTACTS AND LOCATIONS:
Overall Officials: Marieke L Duiverman, Dr, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands